CLINICAL TRIAL: NCT05134779
Title: De-convoluting Interactions Between Genes, the Cancer Environment, and the Immune System to Develop Therapies That Work for You
Acronym: DIGNITY
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 21-06023682
Record Dates: First submitted 2021-10-04; First posted 2021-11-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue collection through the DIGNITY trial will allow the investigators to study the individual tumor and its microenvironment from a biopsy specimen at sequential inflection points and to perform functional genomics experiments using the PDOs technology to determine if the cancer cells can be reprogrammed using radiotherapy and other interventions. Paired blood samples from the patients at each time point will be collected to study circulating cytokines/chemokines, tumor-specific T cells, and innate immune cell response to the PDO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with breast cancer (BC), any stage will be considered for this study.
  Interventions: Procedure: Live Biobank

INTERVENTIONS:
Procedure: Live Biobank — Tumor tissue will be collected from consented patients at sequential inflection points in the disease course: at the time of initial diagnosis, at the time of surgery and during recurrence or metastasis. In addition to this, 40ml of research bloods will also be collected at these key inflection points.

SUMMARY:
This is a live biobank study for breast cancer (BC) patients where samples will be collected at inflection points in the course of the disease.

DETAILED DESCRIPTION:
To test this hypothesis the investigators will focus on studying BC patients using an innovative approach, the DIGNITY Study (De-convoluting interactions between genes, the cancer environment, and the immune system to develop therapies that work for you) designed to building a live tissue biobank of Patient Derived Tumor Organoids (PDOs) derived from tumor at surgery, preceded or not by neoadjuvant therapy (NAT), and at recurrence/metastasis. BC patients enrolled in this study are consented to enable investigators to generate a biobank of tumor tissue (obtained from surgically removed excess that would otherwise be disposed off ) and matched blood cells ( obtained from an already existing line or a venipuncture ordered per standard of care testing) at key timepoints in their treatment course.

ELIGIBILITY:
Inclusion Criteria:

* All patients will historically proven BC are eligible to be on the study

Exclusion Criteria:

* Carriers of other cancers other than breast.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: breast cancer patients (BC), any stage irrespective of hormonal status will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
establish a live biobank for breast cancer patients | 60 months
  Tumor tissue will be obtained at key inflection points from breast cancer patients (BC): at initial diagnosis, at surgery and at metastasis or recurrence.
  Patient Derived Organoids (PDOs) will be prepared from tumors that are obtained from the BC patients.

SECONDARY OUTCOMES:
assess immune relevant genes from tumor biopsies | 60 months
  comprehensively characterize the tumor from the biospecimen to determine the mutations, expression of immune related genes, and the quality and the spatial distribution of the immune infiltrate

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York
  - New York Presbyterian Hospital - Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No